CLINICAL TRIAL: NCT01192581
Title: Hydroxyethyl Starch 130/0.4 and Sodium Chloride Injection as Adjunctive Therapy in Subjects With Internal Carotid Artery Hypoperfusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: the neurology department of Xijing Hospital, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vuloven001
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-06

CONDITIONS: Brain Hypoperfusion
Keywords: brain hypoperfusion; Vuloven; computed tomography perfusion
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (No Intervention): routine treatment for brain hypoperfusion
- Vuloven1 (Experimental): routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 500mg
  Interventions: Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection
- Vuloven2 (Experimental): routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 1000mg
  Interventions: Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection
- Vuloven3 (Experimental): routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 1500mg
  Interventions: Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection

INTERVENTIONS:
Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection — routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 500mg
  Arms: Vuloven1
Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection — routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 1000mg
  Arms: Vuloven2
Drug: hydroxyethyl starch 130/0.4 and sodium chloride injection — routine treatment for brain hypoperfusion plus hydroxyethyl starch 130/0.4 and sodium chloride injection 1500mg
  Arms: Vuloven3

SUMMARY:
The aim of this study is to evaluate the effectiveness, safety and tolerability of consistent dosages of the study drug (hydroxyethyl starch 130/0.4 and sodium chloride injection, Vuloven) administrated intravenously for 7 days.

DETAILED DESCRIPTION:
This study will recruit 120 male and female patients between 18 and 75 years of age who are diagnosed with brain hypoperfusion within the unilateral arteries branching from the internal carotid artery with or without cerebral infarction. All subjects are taking up to routine treatment medications.

The purpose of the study is to evaluate the effectiveness, safety and tolerability of consistent dosages of the study drug (hydroxyethyl starch 130/0.4 and sodium chloride injection, Vuloven) administrated intravenously for 7 days.

Each patient who qualifies and chooses to participate in the study will be randomly assigned into treatment groups (consistent dose of hydroxyethyl starch 130/0.4 and sodium chloride injection of 500 ml/day, 1000 ml/day or 1500 ml/day) or control group (placebo control).

The parameters of clinic visits will include a medical history, physical exam, clinical laboratory tests, magnetic resonance imaging (MRI), using T1-weighted scan, T2-weighted scan and diffusion-weighted imaging (DWI), digital subtraction angiography (DSA), and computed tomography (CT) perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. The degree of the branching arteries stenosis from the internal carotid artery is greater or equal to 70% confirmed by DSA.
2. Before hydroxyethyl starch 130/0.4 and sodium chloride injection-additional treatment, CT perfusion shows that time to peak (TTP) in lesion area is more than that in corresponding area of contralateral hemisphere.
3. If cerebral infarction appears, the time course should be less than 48h, NIH stroke scale: 3-20, and MRI+DWI shows ischemic stroke due to large artery atherosclerosis.

Exclusion Criteria:

1. Allergy to the components of Hydroxyethyl Starch
2. Chronic liver disease (ALT > 120 or AST > 120)
3. Chronic renal disease (Scr > 150 μmol/L)
4. Severe heart failure which correspond to NYHA heart failure classification class III or IV, or serious arrhythmia, myocardial infarction
5. Hemorrhagic stroke
6. Pregnant and lactating women
7. Patients suffered from epilepsy or mental sickness
8. Alcoholism or drug abuse
9. hydroxyethyl starch or other artificial colloidal solution was used within 3 months.
10. Patients participate in other clinical trial within 6 months
11. Contraindication to CT perfusion imaging (i.e. contrast allergy, metformin use or Creatinine >160 μmol/l)
12. Thrombus in lower limb vein

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-04 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy is evaluated based on the measure of CT perfusion parameters | 7 days
  Efficacy is evaluated based on the measure of CT perfusion parameters

SECONDARY OUTCOMES:
Efficacy is evaluated based on scores on NIHSS, Bathl and modified Rankin Scales | 7 days
  Efficacy is evaluated based on scores on NIHSS, Bathl and modified Rankin Scales in those with cerebral infarction
Safety of hydroxyethyl starch 130/0.4 and sodium chloride injection | 7 days
  Safety of hydroxyethyl starch 130/0.4 and sodium chloride injection was evaluated with the monitoring of adverse events (AEs), vital signs, and clinical laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital; Junliang Han, MD, Principal Investigator — Department of Neurology, Xijing Hospital; Fang Yang, MD, PhD, Principal Investigator — Department of Neurology , Xijing Hospital
Locations (1):
- Department of Neurology , Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Han J, Yang F, Jiang W, Zhang G, Liu Z, Liu X, Xia F, Bai Y, He J, Chao M, Zhao G. Hydroxyethyl starch 130/0.4 and sodium chloride injection as adjunctive therapy in patients with cerebral hypoperfusion. BMC Neurol. 2012 Oct 30;12:127. doi: 10.1186/1471-2377-12-127. PMID 23110412